CLINICAL TRIAL: NCT05439213
Title: Comparison of the Effects of Two Concentrations of Adrenaline (0.33 mg/l vs 1 mg/l) in the Irrigation Serum of Arthroscopic Shoulder Surgery.
Acronym: PINHAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GCS Ramsay Santé pour l'Enseignement et la Recherche (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2021-A02773-38
Record Dates: First submitted 2022-06-22; First posted 2022-06-30 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Shoulder Rotator Cuff Tendinitis
MeSH Terms: interventions — Injections; Epinephrine; Solutions

STUDY DESIGN:
Intervention Model Description: Randomised, double-blind, prospective, multicentre study in two parallel groups of 85 patients comparing two concentrations of adrenaline in arthroscopic irrigation fluid (0.33 mg/L vs 1 mg/L
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): adrenaline 0,33 mg per litter
  Interventions: Drug: Adrenaline 0,33 Mg/mL Solution for Injection
- Group 2 (Experimental): adrenaline 1 mg per litter
  Interventions: Drug: Adrenaline 1 Mg/mL Solution for Injection

INTERVENTIONS:
Drug: Adrenaline 0,33 Mg/mL Solution for Injection — adrenaline dosage
  Arms: Group 1
Drug: Adrenaline 1 Mg/mL Solution for Injection — adrenaline dosage
  Arms: Group 2

SUMMARY:
The addition of adrenaline to the arthroscopic irrigation serum is used during rotator cuff surgery to limit intraoperative bleeding and ensure a clear view. Two concentrations of adrenaline are commonly used in practice: 1mg/L or 0.33 mg/L.

The aim of this study is to determine which of these two doses provides better clarity of the surgical field with less impact on the patient's cardiovascular parameters.

DETAILED DESCRIPTION:
A prospective, randomised, double-blind, multicentre study in two parallel groups of 85 patients comparing two concentrations of adrenaline in the irrigation fluid of an arthroscopy (0.33 mg/L vs. 1 mg/L):

Maximum duration of patient participation in the study = 1 day.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years of age, having read and signed the consent form for participation in the study after a reflection period (approximately 15 minutes)
* Patient with a rotator cuff pathology (subacromial impingement, long biceps tendinopathy or rotator cuff tendinopathy)
* Patient for whom an arthroscopic surgical indication has been given

Exclusion Criteria:

* Allergy to epinephrine
* History of Takotsubo cardiomyopathy
* Coagulation disorder
* Patient under court protection, guardianship or curatorship
* Patient not affiliated to the French social security system
* Patient participating in another therapeutic protocol
* Breastfeeding woman,
* Pregnant woman or woman of childbearing age without highly effective contraception for the duration of the study (surgically sterile, intrauterine device (> 14 days), hormonal contraception (same dose and formulation for at least 6 months), sexual abstinence. Women of childbearing age, i.e. fertile, are considered to be post-menopausal unless they are permanently infertile or have undergone surgical sterilisation. A post-menopausal condition is defined as the absence of menstruation for 12 months without any other medical cause
* Patient unable to understand informed information and/or give written informed consent: dementia, psychosis, disturbed consciousness, non-French speaking patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 181 (Actual)
Dates: Start 2022-06-16 (Actual); Primary Completion 2023-06-12 (Actual); Study Completion 2023-06-12 (Actual)

PRIMARY OUTCOMES:
Clarity of the arthroscopic surgical field | Day 1
  The primary endpoint is the clarity of the arthroscopic surgical field assessed by the investigator at the end of the surgical procedure on a numerical scale of 0 to 10, where zero means total opacity throughout the procedure and ten means total clarity throughout the procedure.)

SECONDARY OUTCOMES:
Average blood pressure | Day 1
  The mean intraoperative blood pressure is the average of all measurements taken during the procedure.
Average heart rate | Day 1
  The mean intraoperative heart rate is the average of all measurements taken during the procedure.
Significant changes in blood pressure | Day 1
  The analysis will compare the number of significant changes that occurred in each group and the number of patients per group with at least one significant change.
Significant changes in heart rate | Day 1
  The analysis will compare the number of significant changes that occurred in each group and the number of patients per group with at least one significant change.
Evolution of the pressures of the arthropump | Day 1
  The criteria considered in the analysis will be: the pressure set at the beginning of the procedure, the maximum pressure reached during the procedure and the number of transient hyperpressures requested during the procedure.
Duration of intervention | Day 1
  The duration of the procedure is defined by the time between the beginning of the incision and the end of the suture.
Amount of saline used for the arthroscopic procedure (in litres) | Day 1
  Amount of saline used for the arthroscopic procedure (in litres)

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique de l'Atlantique, Puilboreau, France

IPD SHARING:
Plan to Share IPD: No